CLINICAL TRIAL: NCT03666247
Title: Mobile Messaging Intervention to Present New HIV Prevention Options for MSM - Randomized Controlled Trial
Brief Title: Mobile Messaging Intervention to Present New HIV Prevention Options for Men Who Have Sex With Men (MSM)
Acronym: MMI4MSM RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Patrick S Sullivan, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00087684; 1U01PS004977 (NIH)
Record Dates: First submitted 2018-09-10; First posted 2018-09-11 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Human Immunodeficiency Virus
Keywords: AIDS; Behavioral Science; Infectious Diseases; Health Promotion; Sexually Transmitted Diseases
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Communicable Diseases; Sexually Transmitted Diseases | interventions — Waiting Lists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HealthMindr Application (Experimental): Participants in this study arm will have access to the mobile messaging platform (HealthMindr) for 3 months.
  Interventions: Behavioral: HealthMindr Application
- Waitlist (Other): Participants in this study arm will not have access to the mobile messaging application during the course of the study. After the Month 9 follow up assessment participants in this study arm will be offered access to HealthMindr.
  Interventions: Behavioral: Waitlist

INTERVENTIONS:
Behavioral: HealthMindr Application — From baseline to 3-month post-test, participants in the intervention arm are granted access and instructed to interact regularly with the HealthMindr messaging platform. The HealthMindr messaging platform delivers messages relevant to both general audiences of sexually-active MSM, as well as messages relevant only to specific subgroups of HIV-positive men, and currently higher and lower risk HIV-negative men. Answers provided during the assessments determine which subset of messages are delivered to app users, with information such as HIV status, changes in self-reported risk behaviors, or other factors that influence the relevance of any given message. The HealthMindr application also offers free condoms, lube, and a HIV and STI testing kits.
  Arms: HealthMindr Application
Behavioral: Waitlist — Participants assigned to the waitlist-control arm will be given a welcome sheet orienting them to the study. The message they view will include the same resources links provided to the intervention arm. The information will cover the importance of testing, links to an online mapping tool about the HIV epidemic in the United States (AIDSVu) and resources to locate HIV testing services and prevention information in their area. No information recommending frequency of testing will be given in the welcome greeting.
  Arms: Waitlist

SUMMARY:
The study will evaluate the use and effectiveness of mobile-messaging platforms as a public health strategy for improving sexual health outcome measures among men who have sex with men (MSM) by determining whether exposure to the message-delivery platform results in improvements in participants' self-reported sexual health and prevention behaviors, beliefs and attitudes. The study will enroll men into a randomized controlled trial. Participants randomized to the messaging intervention will have access to a smartphone-based messaging platform for three months while those assigned to the waitlist group will be offered access to the messaging platform after all follow up is complete. Participants will complete surveys at baseline, after the end of the 3 month intervention, and follow up surveys 6 and 9 months after the baseline survey.

DETAILED DESCRIPTION:
This study aims to evaluate the use and effectiveness of a smartphone-based messaging platform as a public health strategy for improving participants' self-reported sexual health and prevention behaviors, beliefs and attitudes. The study will enroll 1,206 men into a randomized controlled trial. They will be assigned to either the immediate intervention group ("intervention arm") or the waitlist-control group ("waitlist-control arm"). All participants will take an assessment survey at baseline, and the intervention group will be oriented on the installation and use of the messaging app upon randomization to that group. All men in the randomized controlled trial will complete short follow-up surveys at 3-month intervals during the 9-month follow-up period. When the intervention arm activities and assessments have concluded, participants in the waitlist-control arm will then be given the option of accessing to the intervention app and participation in intervention post-test activities.

ELIGIBILITY:
Inclusion Criteria:

* Assigned male at birth
* Current, self-reported gender identity as "Male"
* Aged 18 or over
* Self-reported ability to read and understand English-language
* Resides in the Atlanta, Georgia (GA), New York, New York (NY), or Detroit, Michigan (MI) Metropolitan Statistical Area.
* Self-reported anal sex with a male partner in the past 12 months
* Owns and uses an Android or Apple (iOS) smartphone
* Is included in one of the following risk groups, by self-report:

  * HIV seropositive
  * HIV seronegative at "higher risk" (condomless anal sex and not taking PrEP as prescribed in the past 3 months)
  * HIV seronegative at "lower risk" (no condomless anal sex in the past 3 months, or condomless and sex while taking PrEP as prescribed in the past 3 months)

Exclusion Criteria:

* Currently participating in another HIV prevention research study or program
* Participant's phone or device does not support HealthMindr application
* Tested positive for HIV for the first time in the past 6 months
* Has a plan to move out of the Atlanta, GA, New York, NY or Detroit, MI, Metropolitan Statistical Area within in the next 9 months

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1229 (Actual)
Dates: Start 2018-01-24 (Actual); Primary Completion 2019-12-18 (Actual); Study Completion 2019-12-18 (Actual)

PRIMARY OUTCOMES:
Change in HIV testing | Baseline, Month 3, Month 6, Month 9
  HIV-negative men will be asked if they have received an HIV test (ever for the baseline measure and in the past 3 months for follow up surveys).
Change in engagement in HIV care | Baseline, Month 3, Month 6, Month 9
  HIV-positive men will be asked if they have seen a doctor, nurse, or other health provider for HIV care (ever for the baseline measure and in the past 3 months for follow up surveys).
Change in antiretroviral therapy (ART) uptake | Baseline, Month 3, Month 6, Month 9
  HIV-positive men will be asked if they have ever been prescribed and taken antiretroviral medications to treat HIV.
Change in ART adherence | Baseline, Month 3, Month 6, Month 9
  HIV-positive men currently taking antiretroviral medications to treat HIV will be asked if they have been taking their ART as prescribed in the past 3 months.
Change in engagement in HIV preventative care | Baseline, Month 3, Month 6, Month 9
  HIV-negative men will be asked if they have seen a doctor, nurse, or other health care provider (ever for the baseline measure and in the past 3 months for follow up surveys).
Change in pre-exposure prophylaxis (PrEP) uptake | Baseline, Month 3, Month 6, Month 9
  HIV-negative men will be asked if they are taking PrEP (baseline measure) or if they began taking PrEP in the past 3 months (for follow-up measurements).
Change in PrEP adherence | Baseline, Month 3, Month 6, Month 9
  HIV-negative MSM currently taking PrEP will be asked if they have been taking their PrEP medication as prescribed during the past 3 months.
Change in condom use compliance | Baseline, Month 3, Month 6, Month 9
  Proportion of men reporting 100% condom use (stratified by partner type) during the prior 3 months.
Change in condom use | Baseline, Month 3, Month 6, Month 9
  Participants will be asked if they have had any anal sex in which a condom was not used from start to finish in the past 3 months.
Change in testing for sexually transmitted infections (STIs) | Baseline, Month 3, Month 6, Month 9
  Sexually active participants will be asked if they have been tested for STIs in the past 3 months.

SECONDARY OUTCOMES:
Change in intention to engage in preventive behaviors | Baseline, Month 3, Month 6, Month 9
  Participants will report how likely they are to engage in preventive behaviors (such as taking PrEP or ART and increasing condom use) over the next 3 months. Intention to engage in preventive behaviors will be assessed by 11 questions, designed for this study, which are answered on a scale of 1 to 5 where 1 = "definitely not likely" and 5 = "definitely likely". Summed scores can range from 11 to 55 where higher scores indicate increased intention to engage in healthy activities related to HIV prevention and care.
Change in intention to engage in risky behaviors | Baseline, Month 3, Month 6, Month 9
  Participants will report how likely they are to engage in risky behaviors (such as missing doses of PrEP or ART and not using a condom) over the next 3 months. Intention to engage in risky behaviors will be assessed by 3 questions, designed for this study, which are answered on a scale of 1 to 5 where 1 = "definitely not likely" and 5 = "definitely likely". Summed scores can range from 3 to 15 where higher scores indicate increased intention to engage in risky activities related to HIV prevention and care.
Change in intention to seek information | Baseline, Month 3, Month 6, Month 9
  Participants will report how likely they are to seek out information on HIV prevention during the next 3 months.
Change in intention to seek treatment | Baseline, Month 3, Month 6, Month 9
  Participants will report how likely they are to seek out HIV treatment during the next 3 months.
Change in communication with partner | Baseline, Month 3, Month 6, Month 9
  Participants will be asked if they have talked with their sexual partners about ART or PrEP treatment (depending on HIV status) during the past 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Sullivan, PhD, DVM, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Emory University, Atlanta, Georgia
  - University of Michigan, Detroit, Michigan
  - Emory University, New York, New York

REFERENCES:
- [Derived] Sullivan PS, Stephenson R, Hirshfield S, Mehta CC, Zahn R, Bauermeister JA, Horvath K, Chiasson MA, Gelaude D, Mullin S, Downing MJ Jr, Olansky EJ, Wiatrek S, Rogers EQ, Rosenberg E, Siegler AJ, Mansergh G. Behavioral Efficacy of a Sexual Health Mobile App for Men Who Have Sex With Men: Randomized Controlled Trial of Mobile Messaging for Men. J Med Internet Res. 2022 Feb 2;24(2):e34574. doi: 10.2196/34574. PMID 35025755
- [Derived] Sullivan PS, Zahn RJ, Wiatrek S, Chandler CJ, Hirshfield S, Stephenson R, Bauermeister JA, Chiasson MA, Downing MJ Jr, Gelaude DJ, Siegler AJ, Horvath K, Rogers E, Alas A, Olansky EJ, Saul H, Rosenberg ES, Mansergh G. HIV Prevention Via Mobile Messaging for Men Who Have Sex With Men (M-Cubed): Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2019 Nov 15;8(11):e16439. doi: 10.2196/16439. PMID 31730043